CLINICAL TRIAL: NCT01326130
Title: Implementation of an Integrated Primary Care Network for Prevention and Management of Cardiometabolic Risks (RCM)
Brief Title: Implementation of an Integrated Primary Care Network for Prevention and Management of Cardiometabolic Risks
Acronym: RCM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Public Health Department, Montreal (Other Government)
Collaborators: Health and Social Services Agency, Montreal (Other); Fonds de la Recherche en Santé du Québec (Other Government); Ministere de la Sante et des Services Sociaux (Other)
Responsible Party: Pierre Tousignant, Médecin conseil, Public Health Department, Montréal
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RisqueCardioMetabolique; FRSQ 22425 (Other: Fonds de la recherche en santé du Québec)
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes; Hypertension
Keywords: Integrated care network; Chronic care model; Health services research
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Chronic care management 1 (Active Comparator): Content of chronic care model implemented in territory 1 and level of implementation
  Interventions: Behavioral: Chronic care management 1-6
- Chronic care management 2 (Active Comparator): Content of chronic care model implemented in territory 2 and level of implementation
  Interventions: Behavioral: Chronic care management 1-6
- Chronic care management 3 (Active Comparator): Content of chronic care model implemented in territory 3 and level of implementation
  Interventions: Behavioral: Chronic care management 1-6
- Chronic care management 4 (Active Comparator): Content of chronic care model implemented in territory 4 and level of implementation
  Interventions: Behavioral: Chronic care management 1-6
- Chronic care management 5 (Active Comparator): Content of chronic care model implemented in territory 5 and level of implementation
  Interventions: Behavioral: Chronic care management 1-6
- Chronic care management 6 (Active Comparator): Content of chronic care model implemented in territory 6 and level of implementation
  Interventions: Behavioral: Chronic care management 1-6

INTERVENTIONS:
Behavioral: Chronic care management 1-6 — 1- an interdisciplinary team in an education center working with primary care physicians and offering to referred patients a pre-determined sequence of clinical interventions over a 2-year-period; 2- a program supporting primary care physicians (continuing education, documentation and clinical guidelines, referral system to second line of care); 3- networking between actors insuring clinical information transfer required for efficient patient management.

SUMMARY:
CONTEXTE: L'Agence de la santé et des services sociaux de Montréal (ASSS) invited our research team to evaluate the implementation of an integrated and interdisciplinary primary care network for prevention and management of cardiometabolic risks (diabetes and hypertension) (PCR). The intervention is based on the Chronic Care Model and the development of an integrated services network. PCR is to be implemented in 6 territories of "Centre de santé et de services sociaux (CSSS)". A first application for funding was made to Fonds Pfizer-FRSQ-MSSS for an evaluation that has to be completed in the first 24 month after the beginning of the implementation. This application to the PHSI program at CIHR is complementary and will ensure an evaluation of the sustainability of PCR and of long term effects (40 months after the beginning of the implementation) for patients and for their primary care physicians.

In each CSSS, PCR plans for : 1- an interdisciplinary team in an education center working with primary care physicians and offering to referred patients a pre-determined sequence of clinical interventions over a 2-year-period; 2- a program supporting primary care physicians (continuing education, documentation and clinical guidelines, referral system to second line of care); 3- networking between actors of "Réseau local de services (RLS)" insuring clinical information transfer required for efficient patient management.

OBJECTIVES: 1-evaluate PCR effects according to territory, time and degree of exposure (specifically benefits to registered patients and support to participating primary care physicians); 2- identify the degree of implementation of PCR in each CSSS territory and the related contextual factors; 3- examine the relationship between the effects identified, the degree of implementation of PCR and the related contextual factors; 4- assess the impact of implementing PCR on the strengthening of RLS.

METHODS: The proposed evaluation will be done through a mixed design including two complementary strategies. Using a "quasi-experiment/before-after" design, the first strategy is a quantitative approach looking at the program effects and their variation between territories. This analysis will use data from the PCR clinical database (ex.: HbA1c, BP, lifestyle) and from patient questionnaire inquiring about care experience, utilization of services, chronic care follow-up, self-management and quality of life. Around 3000 patients will be enlisted. A primary care physician questionnaire will enquire about PCR effects on their practice. Using primarily a qualitative and a case study approach, each of the 6 territories being one case, the second strategy will identify the degree of implementation of PCR and the explanatory contextual factors. This analysis with use data obtained from semi-structured interviews with program managers. The results of this analysis will be summarized in a monograph for each territory. According to the type of indicator analyzed, objective 3 will be fulfilled using linear models or longitudinal multilevel models supplemented with an interpretive approach using the information from monographs and discussion groups. The impact of implementing PCR on RLS will be assessed through interviews with key informants.

RESULTS AND EXPECTED IMPACT: Our study will identify the effectiveness of PCR and contextual factors associated with successful implementation and sustainability of PCR. Detailed contextual information will allow application of our results to other environments that have similar context and to other chronic conditions that could benefit from an integrated services network.

KNOWLEDGE TRANSFER: Since decision makers, clinicians and researchers did and will take part in all phases of PRC evaluation (planning, data collection, analysis and interpretation), diffusion of information regarding the program is an integral part of the research process. In addition, results will be presented at local, regional, provincial and national conferences and published in reports and articles widely distributed. More specifically, a regional symposium will be organized to share evaluation results with all CSSS in the region (n=12) and with all our local and regional partners.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic adults with borderline fasting blood sugar or glucose intolerance or treated with diet only or treated with only one medication or treated with multiple medications but with Hb A1c ≤ 8%;
* Adults with blood pressure in office ≥ 140/90 mm Hg (if diabetes present, BP ≥ 130/80 mm Hg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Diabetes and Hypertension control | 24 months after registration
  Biomedical indicators of diabetes (Hb A1c ≤7%) and hypertension (blood pressure ≤ 140/90) control

SECONDARY OUTCOMES:
Effects on patient's behavior | 24 months after registration
  Life-style improvement (physical activity, nutrition, smoking)
Effects on patient's autonomy | 24 months after registration
  Self-care
Effects on patient's health | 24 months after registration
  Quality of live
Effects on follow-up of chronic diseases | 24 months after registration
  Chronic care management
Effects on process of care | 24 months after registration
  Indexes of continuity, accessibility, comprehensiveness and perceived quality of care
Effects on physician practice | 24 months after registration
  Physician perception regarding effects of program on patients, inter-professional collaboration, development of knowledge, management of diabetes and hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Tousignant, MD, Principal Investigator — Public Health Department, Montreal
Locations (1):
- Public Health Department, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Provost S, Pineault R, Tousignant P, Hamel M, Da Silva RB. Evaluation of the implementation of an integrated primary care network for prevention and management of cardiometabolic risk in Montreal. BMC Fam Pract. 2011 Nov 10;12:126. doi: 10.1186/1471-2296-12-126. PMID 22074614